CLINICAL TRIAL: NCT03565887
Title: A Randomized, Double-Masked, Placebo-Controlled Phase 3 Study of the Safety and Efficacy of RVL-1201 in the Treatment of Acquired Blepharoptosis
Brief Title: Study of Safety and Efficacy of RVL-1201 in the Treatment of Blepharoptosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RVL Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RVL-1201-202
Record Dates: First submitted 2018-04-11; First posted 2018-06-21 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Blepharoptosis
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RVL-1201 ophthalmic solution 0.1% (Experimental): RVL-1201 (oxymetazoline hydrochloride) ophthalmic solution 0.1%
  Interventions: Drug: RVL-1201
- Vehicle ophthalmic solution (Placebo Comparator): Vehicle placebo ophthalmic solution
  Interventions: Other: Vehicle ophthalmic solution

INTERVENTIONS:
Drug: RVL-1201 — RVL-1201 ophthalmic solution 0.1%
  Arms: RVL-1201 ophthalmic solution 0.1%
Other: Vehicle ophthalmic solution — Vehicle placebo ophthalmic solution
  Arms: Vehicle ophthalmic solution

SUMMARY:
Phase 3 study to evaluate the safety and efficacy of treatment with RVL-1201 compared to placebo for treatment of blepharoptosis. Eligible subjects will be randomized to one of 2 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female 9 years of age or older
2. Females must not be pregnant or planning to get pregnant and must use acceptable form of contraception
3. Must be able to self-administer study medication
4. Must be able to understand and sign an informed consent form. For minor subjects, the subject's parent or legal guardian must provide permission by signing an ICF on behalf of the subject and the subject should provide assent.

Exclusion Criteria:

1. Congenital ptosis
2. Horner syndrome
3. Myasthenia gravis
4. Mechanical ptosis
5. Previous ptosis surgery
6. Resting heart rate outside the normal range
7. Hypertension with resting diastolic blood pressure
8. Pregnancy or lactation

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Barnet, Dulany Perkins, Phoenix, Arizona
  - Orange County Ophthalmology, Garden Grove, California
  - North Valley Eye, Mission Hills, California
  - Eye Research Foundation, Newport Beach, California
  - Pendelton Eye Center, Oceanside, California
  - North Bay Eye Associates, Petaluma, California
  - Michael Tran, Westminster, California
  - Danbury Eye Physicians, Danbury, Connecticut
  - Hernando Eye Institute, Brooksville, Florida
  - Shettle Eye Research, Largo, Florida
  - West Coast Eye, Lecanto, Florida
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center, Maitland, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - East Florida Eye, Stuart, Florida
  - Coastal Research Associates, Roswell, Georgia
  - Kennar Eye Care, Pittsburg, Kansas
  - Heart of America Eye, Shawnee Mission, Kansas
  - Seidenberg Protzko Eye, Havre de Grace, Maryland
  - Mississippi Eye, Ocean Springs, Mississippi
  - Silverstein Eye, Kansas City, Missouri
  - Comprehensive Eye Care, Washington, Missouri
  - Rochester Ophthalmological, Rochester, New York
  - South Shore Eye, Wantagh, New York
  - CEENTA, Charlotte, North Carolina
  - Cornerstone Eye, High Point, North Carolina
  - Quinn, Foster & Assoc., Athens, Ohio
  - Apex Eye, Cincinnati, Ohio
  - Abrams Eye Center, Cleveland, Ohio
  - Nashville vision Associates, Nashville, Tennessee
  - Round Rock Eye, Austin, Texas
  - Texan Eye / Keystone, Austin, Texas
  - Lake Travis Eye, Lakeway, Texas
  - R&R Research, San Antonio, Texas
  - Medical Center Ophthalmology Assocs - Keystone Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned sample size was approximately 156 subjects, 104 subjects in the RVL-1201 group, and 52 in the Vehicle group, to be enrolled at approximately 30 clinical sites in the U.S.
Groups:
- RVL-1201 Ophthalmic Solution 0.1%: RVL-1201 (oxymetazoline hydrochloride) ophthalmic solution 0.1% One drop each eye once-daily in the morning
- Vehicle Ophthalmic Solution: Vehicle placebo ophthalmic Solution One drop each eye once-daily in the morning
Period: Overall Study
Arm/Group | RVL-1201 Ophthalmic Solution 0.1% | Vehicle Ophthalmic Solution
Started | 109 | 55
Completed | 108 | 53
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population
Groups:
- RVL-1201 Ophthalmic Solution 0.1%: RVL-1201 (oxymetazoline hydrochloride) ophthalmic solution 0.1% One drop each eye QD in the morning
- Vehicle Ophthalmic Solution: Vehicle placebo ophthalmic Solution One drop each eye QD in the morning
- Total: Total of all reporting groups
Arm/Group | RVL-1201 Ophthalmic Solution 0.1% | Vehicle Ophthalmic Solution | Total
Number analyzed (Participants) | 109 | 55 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 46 | 22 | 68
  >=65 years | 63 | 32 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (14.31) | 63.3 (16.51) | 63.5 (15.03)
Age, Customized [Median (Full Range); unit: years] | 67.0 [20 to 92] | 67.0 [14 to 85] | 67.0 [14 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 39 | 116
  Male | 32 | 16 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 6 | 19
  Not Hispanic or Latino | 96 | 49 | 145
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 99 | 50 | 149
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 109 | 55 | 164
Iris Color OD (right eye) [Count of Participants; unit: Participants]
  OD-Blue | 40 | 18 | 58
  OD-Brown | 46 | 18 | 64
  OD-Green | 7 | 3 | 10
  OD-Hazel | 15 | 15 | 30
  OD-Grey | 1 | 1 | 2
Iris Color OS (left eye) [Count of Participants; unit: Participants]
  OS-Blue | 40 | 18 | 58
  OS-Brown | 47 | 18 | 65
  OS-Green | 6 | 3 | 9
  OS-Hazel | 15 | 15 | 30
  OS-Grey | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Number of Points Seen on the Leicester Peripheral Field Test (LPFT) in RVL-1201 Group vs. Vehicle Group
Description: LPFT Total Score is the number of points seen in the top 4 rows on the LPFT. Possible scores range from 0 (no points seen) to 35 (all points seen).
Time Frame: Mean change from Baseline (Day 1, Hour 0) compared with Day 1, (Hour 6), and Day 14 (Hour 2)
Population: Intent-to-Treat (ITT) population: randomized who received at least one dose. Per-Protocol Population (PPP): ITT population with no major protocol deviations (eleven subjects were excluded). ITT analysis was conducted for the primary endpoint, with Last Observation Carried Forward (LOCF) for missing data.
Measure: Mean (Standard Deviation); unit: Points seen
Arm/Group | RVL-1201 Ophthalmic Solution 0.1% | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 109 | 55
Points seen
  Mean change from baseline LPFT-Day 1 Hour 6 | 6.3 (6.72) | 2.1 (4.28)
  Mean change from baseline LPFT-Day 14 Hour 2 | 7.7 (6.41) | 2.4 (5.26)
Statistical Analysis 1: Comparison: RVL-1201 Ophthalmic Solution 0.1% vs Vehicle Ophthalmic Solution; A two group t-test with a 0.05 two-sided significance level had 90% power to detect a difference in LPFT means of 3.50 assuming that the common standard deviation was 6.0, when the sample sizes in the 2 groups were 94 and 47, respectively (a total sample size of 141); Test type: Superiority — The primary efficacy endpoints were tested sequentially. The Day 1 Hour 6 time point was tested first and if P<0.05, the Day 14 Hour 2 time point was tested at a significance level of 0.05. If the Day 1 Hour 6 endpoint is statistically significant (at the 0.05 level) but Day 14 Hour 2 was not statistically significant (at the 0.05 level), the study will still be considered positive; p < 0.0001, ANCOVA — If both primary endpoints (LPFT) are significant at 0.05 significance level, then the secondary efficacy endpoints (MRD) were also tested sequentially. Testing stopped if a P≥ 0.05 for a comparison; 2 sided t-test with treatment as fixed factor and baseline as covariate

2. Secondary Outcome: Mean Change From Baseline in Marginal Reflex Distance (MRD) in the Study Eye
Description: The Marginal Reflex Distance (MRD) is the distance from the center pupillary light reflex to the central margin of the upper eyelid. The MRD is measured from an external photograph using a handheld caliper and a millimeter ruler label placed on the subject's forehead as a measurement legend.
Time Frame: Baseline Day 1 (Hour 0) and Day 1, Day 14, and Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | RVL-1201 Ophthalmic Solution 0.1% | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 109 | 55
Millimeters (mm)
  Day 1, Minute 5 | 0.59 (0.721) | 0.20 (0.571)
  Day 1, Minute 15 | 0.93 (0.811) | 0.32 (0.641)
  Day 1, Hour 2 | 1.05 (0.903) | 0.33 (0.555)
  Day 1, Hour 6 | 0.98 (0.867) | 0.35 (0.567)
  Day 14, Minute 5 | 0.77 (0.853) | 0.42 (0.775)
  Day 14, Minute 15 | 1.11 (0.922) | 0.41 (0.833)
  Day 14, Hour 2 | 1.22 (0.926) | 0.43 (0.734)
  Day 14, Hour 6 | 1.06 (0.902) | 0.47 (0.737)
  Day 42, Minute 5 | 0.86 (0.849) | 0.42 (0.799)
  Day 42, Minute 15 | 1.04 (0.912) | 0.47 (0.926)
Statistical Analysis 1: Comparison: RVL-1201 Ophthalmic Solution 0.1% vs Vehicle Ophthalmic Solution; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — If both primary endpoints (LPFT) are significant at 0.05 significance level, then the secondary efficacy endpoints (MRD) were also tested sequentially. Testing stopped if a P≥ 0.05 for a comparison; p < 0.0151, ANCOVA

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) were assessed at Baseline through Day 42 (end of study).
Description: AEs spontaneously reported by the subject and/or in response to an open questions from the study personnel or revealed by observation were recorded in the eCRF.
Groups:
- RVL-1201 Ophthalmic Solution, 0.1%: One drop each eye QD in the morning (n=109)
- Vehicle Ophthalmic Solution: One drop each eye QD in the morning (n=55)
Arm/Group | RVL-1201 Ophthalmic Solution, 0.1% | Vehicle Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/109 | 1/55
Other Adverse Events (participants affected / at risk) | 13/109 | 8/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RVL-1201 Ophthalmic Solution, 0.1% (N=109) | Vehicle Ophthalmic Solution (N=55)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RVL-1201 Ophthalmic Solution, 0.1% (N=109) | Vehicle Ophthalmic Solution (N=55)
Conjunctival hyperaemia (Eye disorders) | 6 (10) | 1 (2)
Punctate keratitis (Eye disorders) | 4 (8) | 1 (1)
Eye pain (Eye disorders) | 3 (4) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 2 (4)
Instillation site complication (General disorders) | 0 (0) | 2 (4) — Administration site conditions
Vital dye straining cornea present (Investigations) | 1 (2) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT03565887/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT03565887/SAP_001.pdf